CLINICAL TRIAL: NCT02999464
Title: Effect of Qigong on Balance, Fall Efficacy, Physical Functions and Psychological Wellbeing of People With Stroke in Hong Kong: A Randomized Controlled Trial
Brief Title: Effect of Qigong on Balance, Fall Efficacy, Wellbeing of People With Stroke in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Yuen Shuk Man, Principal investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20151013001
Record Dates: First submitted 2016-04-24; First posted 2016-12-21 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
Keywords: stroke; qigong; randomized controlled trial; body-mind exercise; balance; quality of life; wellbeing
MeSH Terms: conditions — Stroke | interventions — Qigong; Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Qigong (Experimental): Experimental group will receive a total of 50 minutes of qigong training 3 times per week and for 16 weeks.
  Interventions: Other: Qigong
- Fitness Exercise (Active Comparator): Fitness exercise group will receive home fitness exercise 3 times per week and for 16 weeks.
  Interventions: Other: Fitness exercise

INTERVENTIONS:
Other: Qigong — The experimental group will be required to practice a total of 50 minutes of qigong training 3 times per week and for 16 weeks
  Other Names: body-mind exercise
  Arms: Qigong
Other: Fitness exercise — Active control group will be required to practice a total of 50 minutes of fitness training 3 times per week and for 16 weeks
  Arms: Fitness Exercise

SUMMARY:
The purpose of this study is to compare the effects of qigong practice with fitness exercise on balance, fall-efficacy, physical functions, psychological wellbeing and quality of life of stroke survivors.

DETAILED DESCRIPTION:
Participants: A total of 58 stroke survivors 3 months after the current stroke will be recruited.

Methodology: An assessor-blinded, randomized controlled trial will be conducted. Stroke survivors will be included in the study if they meet the inclusion criteria. Selected patients will be randomly allocated into either the experimental group or the control group. Participants allocated in the experimental group will receive qigong training while this qigong training will be replaced by a home fitness exercise in the control group. The experimental and control groups will be required to practice a total of 50 minutes of qigong and fitness training 3 times per week and for 16 weeks respectively. The main outcome measure is balance capacity with Mini-BESTest. The secondary outcomes are fall efficacy, number of falls, postural stability and control, depression, physical functions and quality of life. Assessments will be done at baseline, 8 weeks and 16 weeks follow-ups by blinded assessors.

Data analysis: The results will be analyzed using two-way repeated measures analysis of variance with Statistical Package for Social Science version 21.0. Alpha will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke and 3 months after the onset
* First episode of stroke or recurrent of stroke
* Able to stand for more than 15 minutes
* Able to take anterioposterior and lateral step without assistance or aid
* Medically stable
* Sufficient cognition to follow commands Abbreviated Mental Test (AMT) score ≥7

Exclusion Criteria:

* Vital signs unstable
* History or evidence of other neurological deficits other than stroke such as multiple sclerosis
* Severe primary diseases of the cardiovascular system, liver, kidney or hematopoietic system
* Experience in qigong practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Mini-BESTest. | Baseline, 8th week and 16th week after intervention
  Change from baseline balance capacity at 8 weeks and 16 weeks

SECONDARY OUTCOMES:
Fall Efficacy Scale - International | Baseline, 8th week and 16th week after intervention
  Change from baseline fall efficacy of the subject at 8 weeks and 16 weeks
Number of falls | Baseline, 8th week and 16th week after intervention
Limit of Stability by using Balance Master | Baseline, 8th week and 16th week after intervention
  Change from baseline postural stability at 8 weeks and 16 weeks
Geriatric Depression Scale | Baseline, 8th week and 16th week after intervention
Five Times Sit to Stand Test | Baseline, 8th week and 16th week after intervention
  Lower extremity strength
Timed Up and Go Test | Baseline, 8th week and 16th week after intervention
  Change from baseline gait speed at 8 weeks and 16 weeks
Modified Barthel Index | Baseline, 8th week and 16th week after intervention
  Activities of daily living function
Stroke-Specific Quality of Life Scale | Baseline, 8th week and 16th week after intervention
Sensory Organization Test by using Balance Master | Baseline, 8th week and 16th week after intervention
  Change from baseline postural control at 8 weeks and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yiu-chung PANG, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Kowloon Hospital, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yuen M, Ouyang HX, Miller T, Pang MYC. Baduanjin Qigong Improves Balance, Leg Strength, and Mobility in Individuals With Chronic Stroke: A Randomized Controlled Study. Neurorehabil Neural Repair. 2021 May;35(5):444-456. doi: 10.1177/15459683211005020. Epub 2021 Apr 7. PMID 33825587